CLINICAL TRIAL: NCT02614729
Title: A Randomized Controlled Feeding, Crossover Trial to Assess the Appetitive and Cognitive Effects of Daily Beef Consumption in Healthy, Overweight Women
Brief Title: The Consumption of Beef on Appetite and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, Heather Leidy, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 0039674
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Obesity; Poor Glycemic Control; Dietary Interventions
Keywords: High Protein; Satiety; Appetite Control; Protein Distribution; Cognitive Function; Ad libitum Food Intake; Obesity prevention; Obesity treatment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy Balance Comparison (Experimental): Participants will randomly consume 4 eucaloric diets for 7 consecutive days/treatment. Energy levels for all diets are established according to needs for energy balance.
  Interventions:
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN); Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN); High Protein-Beef, Even Distribution (HP-BEEF-EVEN); High Protein-Beef, Uneven Distribution (HP-BEEF-UNEVEN)
  Interventions: Other: Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN); Other: Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN); Other: High Protein-Beef, Even Distribution (HP-BEEF-EVEN); Other: High Protein-Beef, Uneven Distribution (HP-BEEF-UNEVEN)
- Energy Restriction Comparison (Experimental): Participants will randomly consume 3 energy restriction diets (1250 kcal/day) for 7 consecutive days/treatment. Energy levels for all diets are established according to needs for energy restriction.
  Interventions:
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN); Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN); High Protein-Beef, Even Distribution (HP-BEEF-EVEN)
  Interventions: Other: Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN); Other: Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN); Other: High Protein-Beef, Even Distribution (HP-BEEF-EVEN)

INTERVENTIONS:
Other: Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN) — Diet contains all plant proteins. Meals are evenly distributed throughout the day.
Other: Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN) — Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
Other: High Protein-Beef, Even Distribution (HP-BEEF-EVEN) — Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
Other: High Protein-Beef, Uneven Distribution (HP-BEEF-UNEVEN) — Diet contains combination of beef and plant proteins. Meals are unevenly distributed throughout the day.
  Arms: Energy Balance Comparison

SUMMARY:
The purpose of the main study is to determine whether the daily consumption of protein-rich meals containing high quality, lean beef products improves appetite control and cognitive function during a weight maintenance diet.

The purpose of the sub-study is to determine whether the daily consumption of protein-rich meals containing the same amount of high quality, lean beef products improves appetite control and cognitive function during a modest energy restriction, weight loss diet.

DETAILED DESCRIPTION:
Two cross-over design studies were completed in overweight, sedentary but otherwise healthy women. For study 1, 17 participants randomly consumed 4 eucaloric diets containing standard-protein (SP; 76±1g protein/d) or high-protein (HP; 126±1g protein/d) for 7 consecutive days/treatment. The SP treatments contained all plant proteins (PLANT) or a combination of beef and plant proteins (BEEF) that were evenly distributed throughout the day (EVEN). The HP treatments were also BEEF provided as EVEN or an uneven distribution (UNEVEN) pattern. For study 2, 17 participants randomly consumed 3 energy restriction (1250 kcal/d) diets containing SP-PLANT (EVEN) and SP-BEEF (EVEN) (both, 48±1g protein/d) or HP-BEEF (EVEN) (123±1g protein/d). During day 6 of each treatment (for both studies), the participants completed a 12-h controlled-feeding, clinical testing day which included repeated appetite, satiety, food cravings, and mood questionnaires; blood sampling; and cognitive function/performance testing. During day 7 of each treatment (for both studies), the participants completed a free-living, ad libitum testing day at home/work to assess ad libitum (voluntary) daily intake and food choice. Each of the 7-day dietary patterns occurred during the follicular phase of the menstrual cycle; thus, there were 2-3 week washout periods between dietary treatments.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Ages: 18-52 y
* BMI: 25-32 kg/m2
* No metabolic, hormonal, and/or neural conditions/diseases that influence metabolism, appetite, or cognition
* No blood donations to American Red Cross within past 6 months
* No medication that would influence directly appetite or cognition
* No change in any medications (over the past 3 months)
* Non-smoking (for the past year)
* Not pregnant within the past 6 months (or planning to become pregnant during study)
* Have not given birth and/or lactating within the past 6 months
* Normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or able to provide documentation of oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos)
* Not clinically diagnosed with an eating disorder
* No weight loss/gain (≥10 lb. in the past 6 months)
* No past history of surgical interventions for the treatment of obesity
* No allergies and/or aversions to the study foods, particularly beef
* Consumes ≤ 800 mg caffeine/day
* Of this, ≤260 mg caffeine is consumed prior to lunch (~12 oz. Starbucks coffee)
* Not currently and/or previously on a specific diet including high protein, vegan, vegetarian, etc.
* Willing and able to consume all study foods
* Habitually consumes breakfast, lunch, and dinner >4 days/week
* No history of drug abuse or alcohol abuse (i.e., >14 drinks/week; 1 drink=12 oz. beer; 5 oz. wine; 1.5 oz. liquor)
* Displays a score of <4 on the Three Factor Eating Habits Questionnaire (TFEQ)
* Conventional (typical) and consistent sleep patterns
* awake hours somewhere between 5 am - 11 pm with no afternoon naps
* rates quality of sleep as Fairly to Very Good on the Pittsburg Sleep Quality Index (PSQI)
* averages ≥ 6 sleep hours/night over the past month
* Displays a Profile of Mood State 2nd Edition (POMS2; 60-item) Depression-Dejection Scale score within 1.5 SD of the age, gender, and racial-specific normative mean (Nyenhuis et al., 1999; Petterson K et al., 2006)
* Obtained a "Yes" on the validity indicator and displayed a score of >70 (>2%) on the CNS Vital Signs Battery
* Sedentary (i.e., limited purposeful physical activity)
* Willing and able to maintain current inactivity patterns throughout the study
* Willing and able to follow all study procedures
* Generally healthy, as assessed from the medical history questionnaire

Exclusion Criteria:

* Men
* Ages: <18 or >52 y
* BMI: <25 or >32 kg/m2
* Any metabolic, hormonal, and/or neural conditions/diseases that influence metabolism, appetite, or cognition
* Have donated blood to American Red Cross within past 6 months
* Medication that would influence directly appetite or cognition
* Change in medications (over the past 3 months)
* Have smoked in the past year
* Pregnant within the past 6 months (or planning to become pregnant during study)
* Have given birth and/or lactating within the past 6 months
* Abnormal menstrual cycles [not between 26-32 days in duration; or not 5-6 menstrual cycles within the past 6 months; or not able to provide documentation of oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos)]
* Clinically diagnosed with an eating disorder
* Weight loss/gain (≥10 lb. in the past 6 months)
* Past history of surgical interventions for the treatment of obesity
* Allergies and/or aversions to the study foods, particularly beef
* Consumes > 800 mg caffeine/day
* Or, of caffeine consumed, >260 mg caffeine is consumed prior to lunch (~12 oz. Starbucks coffee)
* Currently and/or previously on a specific diet including high protein, vegan, vegetarian, etc.
* Unwilling and/or unable to consume all study foods
* Habitually consumes breakfast, lunch, and dinner <4 days/week
* History of drug abuse or alcohol abuse (i.e., >14 drinks/week; 1 drink=12 oz. beer; 5 oz. wine; 1.5 oz. liquor)
* Displays a score of >4 on the Three Factor Eating Habits Questionnaire (TFEQ)
* Unconventional (atypical) and/or inconsistent sleep patterns
* awake hours not somewhere between 5 am - 11 pm and/or afternoon naps
* does not rate quality of sleep as Fairly to Very Good on the Pittsburg Sleep Quality Index (PSQI)
* averages < 6 sleep hours/night over the past month
* Does not display a Profile of Mood State 2nd Edition (POMS2; 60-item) Depression-Dejection Scale score within 1.5 SD of the age, gender, and racial-specific normative mean (Nyenhuis et al., 1999; Petterson K et al., 2006)
* Did not obtain a "Yes" on the validity indicator and/or did not display a score of >70 (>2%) on the CNS Vital Signs Battery
* Not sedentary (i.e., purposeful physical activity)
* Unwilling and/or unable to maintain current inactivity patterns throughout the study
* Unwilling and/or unable to follow all study procedures
* Not generally healthy, as assessed from the medical history questionnaire

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leidy HJ, Clifton PM, Astrup A, Wycherley TP, Westerterp-Plantenga MS, Luscombe-Marsh ND, Woods SC, Mattes RD. The role of protein in weight loss and maintenance. Am J Clin Nutr. 2015 Jun;101(6):1320S-1329S. doi: 10.3945/ajcn.114.084038. Epub 2015 Apr 29. PMID 25926512
- [Background] Holt SH, Miller JC, Petocz P, Farmakalidis E. A satiety index of common foods. Eur J Clin Nutr. 1995 Sep;49(9):675-90. PMID 7498104
- [Background] Leidy HJ, Carnell NS, Mattes RD, Campbell WW. Higher protein intake preserves lean mass and satiety with weight loss in pre-obese and obese women. Obesity (Silver Spring). 2007 Feb;15(2):421-9. doi: 10.1038/oby.2007.531. PMID 17299116
- [Background] Layman DK, Boileau RA, Erickson DJ, Painter JE, Shiue H, Sather C, Christou DD. A reduced ratio of dietary carbohydrate to protein improves body composition and blood lipid profiles during weight loss in adult women. J Nutr. 2003 Feb;133(2):411-7. doi: 10.1093/jn/133.2.411. PMID 12566476
- [Background] Johnston CS, Tjonn SL, Swan PD. High-protein, low-fat diets are effective for weight loss and favorably alter biomarkers in healthy adults. J Nutr. 2004 Mar;134(3):586-91. doi: 10.1093/jn/134.3.586. PMID 14988451
- [Background] Mamerow MM, Mettler JA, English KL, Casperson SL, Arentson-Lantz E, Sheffield-Moore M, Layman DK, Paddon-Jones D. Dietary protein distribution positively influences 24-h muscle protein synthesis in healthy adults. J Nutr. 2014 Jun;144(6):876-80. doi: 10.3945/jn.113.185280. Epub 2014 Jan 29. PMID 24477298
- [Background] Leidy HJ, Bossingham MJ, Mattes RD, Campbell WW. Increased dietary protein consumed at breakfast leads to an initial and sustained feeling of fullness during energy restriction compared to other meal times. Br J Nutr. 2009 Mar;101(6):798-803. doi: 10.1017/s0007114508051532. PMID 19283886
- [Background] Hoyland A, Dye L, Lawton CL. A systematic review of the effect of breakfast on the cognitive performance of children and adolescents. Nutr Res Rev. 2009 Dec;22(2):220-43. doi: 10.1017/S0954422409990175. PMID 19930787
- [Background] Benau EM, Orloff NC, Janke EA, Serpell L, Timko CA. A systematic review of the effects of experimental fasting on cognition. Appetite. 2014 Jun;77:52-61. doi: 10.1016/j.appet.2014.02.014. Epub 2014 Feb 27. PMID 24583414
- [Background] Spring B, Maller O, Wurtman J, Digman L, Cozolino L. Effects of protein and carbohydrate meals on mood and performance: interactions with sex and age. J Psychiatr Res. 1982-1983;17(2):155-67. doi: 10.1016/0022-3956(82)90017-6. PMID 6764932
- [Background] Jakobsen LH, Kondrup J, Zellner M, Tetens I, Roth E. Effect of a high protein meat diet on muscle and cognitive functions: a randomised controlled dietary intervention trial in healthy men. Clin Nutr. 2011 Jun;30(3):303-11. doi: 10.1016/j.clnu.2010.12.010. Epub 2011 Jan 15. PMID 21239090
- [Background] Lieberman HR, Spring BJ, Garfield GS. The behavioral effects of food constituents: strategies used in studies of amino acids, protein, carbohydrate and caffeine. Nutr Rev. 1986 May;44 Suppl:61-70. doi: 10.1111/j.1753-4887.1986.tb07679.x. No abstract available. PMID 2980858
- [Background] Finnigan F, Hammersley R, Millar K. Effects of meal composition on blood alcohol level, psychomotor performance and subjective state after ingestion of alcohol. Appetite. 1998 Dec;31(3):361-75. doi: 10.1006/appe.1998.0168. PMID 9920688
- [Background] Nyenhuis DL, Yamamoto C, Luchetta T, Terrien A, Parmentier A. Adult and geriatric normative data and validation of the profile of mood states. J Clin Psychol. 1999 Jan;55(1):79-86. doi: 10.1002/(sici)1097-4679(199901)55:13.0.co;2-7. PMID 10100834
- [Background] Patterson K, Young C, Woods SP, Vigil O, Grant I, Atkinson JH; HIV Neurobehavioral Research Center Group. Screening for major depression in persons with HIV infection: the concurrent predictive validity of the Profile of Mood States Depression-Dejection Scale. Int J Methods Psychiatr Res. 2006 Jun;15(2):75-82. doi: 10.1002/mpr.184. PMID 19722288
- [Background] Paddon-Jones D, Leidy H. Dietary protein and muscle in older persons. Curr Opin Clin Nutr Metab Care. 2014 Jan;17(1):5-11. doi: 10.1097/MCO.0000000000000011. PMID 24310053
- [Background] White MA, Whisenhunt BL, Williamson DA, Greenway FL, Netemeyer RG. Development and validation of the food-craving inventory. Obes Res. 2002 Feb;10(2):107-14. doi: 10.1038/oby.2002.17. PMID 11836456
- [Background] Gualtieri CT, Johnson LG. Reliability and validity of a computerized neurocognitive test battery, CNS Vital Signs. Arch Clin Neuropsychol. 2006 Oct;21(7):623-43. doi: 10.1016/j.acn.2006.05.007. Epub 2006 Oct 2. PMID 17014981
- [Background] Leidy HJ, Tang M, Armstrong CL, Martin CB, Campbell WW. The effects of consuming frequent, higher protein meals on appetite and satiety during weight loss in overweight/obese men. Obesity (Silver Spring). 2011 Apr;19(4):818-24. doi: 10.1038/oby.2010.203. Epub 2010 Sep 16. PMID 20847729
- [Background] Leidy HJ, Armstrong CL, Tang M, Mattes RD, Campbell WW. The influence of higher protein intake and greater eating frequency on appetite control in overweight and obese men. Obesity (Silver Spring). 2010 Sep;18(9):1725-32. doi: 10.1038/oby.2010.45. Epub 2010 Mar 25. PMID 20339363
- [Background] Weigle DS, Breen PA, Matthys CC, Callahan HS, Meeuws KE, Burden VR, Purnell JQ. A high-protein diet induces sustained reductions in appetite, ad libitum caloric intake, and body weight despite compensatory changes in diurnal plasma leptin and ghrelin concentrations. Am J Clin Nutr. 2005 Jul;82(1):41-8. doi: 10.1093/ajcn.82.1.41. PMID 16002798
- [Background] Leidy HJ, Todd CB, Zino AZ, Immel JE, Mukherjea R, Shafer RS, Ortinau LC, Braun M. Consuming High-Protein Soy Snacks Affects Appetite Control, Satiety, and Diet Quality in Young People and Influences Select Aspects of Mood and Cognition. J Nutr. 2015 Jul;145(7):1614-22. doi: 10.3945/jn.115.212092. Epub 2015 May 20. PMID 25995282
- [Background] Zeng YC, Li SM, Xiong GL, Su HM, Wan JC. Influences of protein to energy ratios in breakfast on mood, alertness and attention in the healthy undergraduate students. Health 3(6): 383-393. 2011
- [Background] Russell JA. Affect Grid: A single-item scale of pleasure and arousal. J Personality Soc Psychol 57 (3): 493-502, 1989.
- [Derived] Piacquadio KA, Gwin JA, Leidy HJ. A Higher-Protein, Energy Restriction Diet Containing 4 Servings of Fresh, Lean Beef per Day Does Not Negatively Influence Circulating miRNAs Associated with Cardiometabolic Disease Risk in Women with Overweight. Curr Dev Nutr. 2024 Aug 18;8(9):104442. doi: 10.1016/j.cdnut.2024.104442. eCollection 2024 Sep. PMID 39310667
- [Derived] Braden ML, Gwin JA, Leidy HJ. A Diet Containing Animal Source Protein as Fresh, Lean Beef Is More Well Liked and Promotes Healthier Eating Behavior Compared with Plant-Based Alternatives in Women with Overweight. Curr Dev Nutr. 2024 Jul 14;8(8):104415. doi: 10.1016/j.cdnut.2024.104415. eCollection 2024 Aug. PMID 39224138
- [Derived] Piacquadio KA, Margolis LM, Gwin JA, Leidy HJ. Higher Expression of miR-15b-5p with Inclusion of Fresh, Lean Beef as Part of a Healthy Dietary Pattern Is Inversely Associated with Markers of Cardiometabolic Disease Risk. J Nutr. 2024 Jun;154(6):1758-1765. doi: 10.1016/j.tjnut.2024.04.026. Epub 2024 Apr 25. PMID 38677478
- [Derived] Gwin JA, Maki KC, Alwattar AY, Leidy HJ. Examination of Protein Quantity and Protein Distribution across the Day on Ad Libitum Carbohydrate and Fat Intake in Overweight Women. Curr Dev Nutr. 2017 Oct 25;1(12):e001933. doi: 10.3945/cdn.117.001933. eCollection 2017 Dec. PMID 29955692
- [Derived] Gwin JA, Maki KC, Leidy HJ. Increased Protein Consumption during the Day from an Energy-Restricted Diet Augments Satiety but Does Not Reduce Daily Fat or Carbohydrate Intake on a Free-Living Test Day in Overweight Women. J Nutr. 2017 Dec;147(12):2338-2346. doi: 10.3945/jn.117.255554. Epub 2017 Oct 25. PMID 29070709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from Columbia, Missouri and the surrounding area from January 2014 to May 2015.
Pre-assignment Details: Following recruitment and screening, 17 met women met the screening criteria, signed the study consent, and completed the study procedures. All participants received the following treatments: Energy Balance Comparison (n=17) (SP-PLANT, SP-BEEF, HP-BEEF-EVEN, HP-BEEF-SKEW) & Energy Restriction Comparison (n=17) (SP-PLANT, SP-BEEF, HP-BEEF-EVEN).
Groups:
- Energy Balance Comparison: Participants will randomly consume 4 eucaloric diets for 7 consecutive days/treatment. Energy levels for all diets are established according to needs for energy balance.
  Interventions:
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN); Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN); High Protein-Beef, Even Distribution (HP-BEEF-EVEN); High Protein-Beef, Uneven Distribution (HP-BEEF-UNEVEN)
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN): Diet contains all plant proteins. Meals are evenly distributed throughout the day.
  Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN): Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
  High Protein-Beef, Even Distribution (HP-BEEF-EVEN): Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
  High Protein-Beef, Uneven Distribution (HP-BEEF-UNEVEN): Diet contains combination of beef and plant proteins. Meals
- Energy Restriction Comparison: Participants will randomly consume 3 energy restriction diets (1250 kcal/day) for 7 consecutive days/treatment. Energy levels for all diets are established according to needs for energy restriction.
  Interventions:
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN); Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN); High Protein-Beef, Even Distribution (HP-BEEF-EVEN)
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN): Diet contains all plant proteins. Meals are evenly distributed throughout the day.
  Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN): Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
  High Protein-Beef, Even Distribution (HP-BEEF-EVEN): Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
Period: Overall Study
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Daily Energy Intake: Total Daily Intake
Description: Energy intake during breakfast, lunch, dinner, and evening snacks of each day 7 testing day (separated by 3-4 weeks) will be measured.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: kcal
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
kcal
  SP-PLANT | 2859 (147) | 2313 (170)
  SP-BEEF | 2714 (219) | 2396 (181)
  HP-BEEF-EVEN | 2830 (214) | 2820 (173)
  HP-BEEF-SKEW | 3039 (184) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

2. Secondary Outcome: Perceived Fullness
Description: Questionnaires assessing fullness will be completed throughout each of the 12-hour testing days (which are separated by 3-4 weeks). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The scale is 0 to 100mm. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not at all" (indicated at 0 mm) to "extremely" (indicated at 100 mm). All measures are reported at area under the curve for 0 to 630 min.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: Total Fullness AUC (mm*630 min)
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
Total Fullness AUC (mm*630 min)
  SP-PLANT: Daily Fullness | 38849 (2302) | 32167 (2745)
  SP-BEEF: Daily Fullness | 38689 (2235) | 30862 (2896)
  HP-BEEF-EVEN: Daily Fullness | 39560 (2536) | 36313 (2260)
  HP-BEEF-SKEW: Daily Fullness | 38464 (2693) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

3. Secondary Outcome: Reaction Time as a Measure of Cognitive Performance Assessed Using the Stroop Test
Description: Cognitive function will be assessed during each of the 12-hour testing days using CNS Vital Signs, a validated computerized assessment. This system contains a core battery of tasks. Reaction Time is the outcome of interest measured with the Stroop Test. In the first part, the words RED, YELLOW, BLUE, & GREEN (printed in black) appear at random on the screen, & the participant presses the space bar as soon as the test subject sees the word. In the second part, the words RED, YELLOW, BLUE, & GREEN appear on the screen, printed in color. The participant is asked to press the space bar when the color of the word matches what the word says. In the third part, the words RED, YELLOW, BLUE, & GREEN appear on the screen, printed in color. The participant is asked to press the space bar when the color of the word does not match what the word says. Reaction time is in milliseconds.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: ms
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
ms
  SP-PLANT: Reaction Time | 309 (7) | 303 (8)
  SP-BEEF: Reaction Time | 321 (7) | 311 (6)
  HP-BEEF-EVEN: Reaction Time | 320 (9) | 312 (7)
  HP-BEEF-SKEW: Reaction Time | 317 (9) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

4. Secondary Outcome: Perceived Alertness
Description: Alertness will be assessed during each of the 12-hour testing days (which are separated by 3-4 weeks) using the Profile of Mood States 2nd Edition (POMS2) with sub-categories of perceived vigor. POM2 is a self-report measure that allows for the quick assessment of transient, fluctuating feelings, and enduring affect states. There are 35 items. Items are rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The Alertness (Vigor-Activity) scale score indicates the extent to which individual felt alert (vigorous and/or energetic); the higher are her positive feelings and/or energy, the greater is her score (i.e., a low score indicates relatively fewer positive feelings and/or low energy). Ratings on this scale yielded a T-score of 25 (95% CI =18-32), which is ranked at the 1st percentile, and falls within the Very Low score range. The T scores were then used to calculate area under the curve.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: Total AUC (T-score*min)
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
Total AUC (T-score*min)
  SP-PLANT: Total Alertness | 1631 (448) | 2151 (883)
  SP-BEEF: Total Alertness | 1525 (638) | 1950 (631)
  HP-BEEF-EVEN: Total Alertness | 1374 (424) | 2434 (954)
  HP-BEEF-SKEW: Total Alertness | 1414 (712) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

5. Secondary Outcome: Perceived Hunger
Description: Questionnaires assessing hunger will be completed throughout each of the 12-hour testing days (which are separated by 3-4 weeks). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The scale is 0 to 100mm. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not at all" (indicated at 0 mm) to "extremely" (indicated at 100 mm). All measures are reported at area under the curve for 0 to 630 min.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: Total Fullness AUC (mm*630 min)
Groups:
- Energy Balance Comparison: Participants will randomly consume 4 eucaloric diets for 7 consecutive days/treatment. Energy levels for all diets are established according to needs for energy balance.
  Interventions:
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN): Diet contains all plant proteins. Meals are evenly distributed throughout the day.
  Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN): Diet contains combination of beef & plant proteins. Meals are evenly distributed throughout the day.
  High Protein-Beef, Even Distribution (HP-BEEF-EVEN): Diet contains combination of beef & plant proteins. Meals are evenly distributed throughout the day.
  High Protein-Beef, Uneven Distribution (HP-BEEF-UNEVEN): Diet contains combination of beef & plant proteins. Meals are unevenly distributed throughout the day.
- Energy Restriction Comparison: Participants will randomly consume 3 energy restriction diets (1250 kcal/day) for 7 consecutive days/treatment. Energy levels for all diets are established according to needs for energy restriction.
  Interventions:
  Standard Protein-Plant, Even Distribution (SP-PLANT-EVEN): Diet contains all plant proteins. Meals are evenly distributed throughout the day.
  Standard Protein-Beef, Even Distribution (SP-BEEF-EVEN): Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
  High Protein-Beef, Even Distribution (HP-BEEF-EVEN): Diet contains combination of beef and plant proteins. Meals are evenly distributed throughout the day.
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
Total Fullness AUC (mm*630 min)
  SP-PLANT: Daily Hunger | 16624 (1989) | 21833 (2370)
  SP-BEEF: Daily Hunger | 17496 (1836) | 24849 (2557)
  HP-BEEF-EVEN: Daily Hunger | 16713 (1831) | 18598 (1868)
  HP-BEEF-SKEW: Daily Hunger | 17689 (1829) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

6. Secondary Outcome: Perceived Prospective Food Consumption
Description: Questionnaires assessing prospective food consumption will be completed throughout each of the 12-hour testing days (which are separated by 3-4 weeks). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The scale is 0 to 100mm. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not at all" (indicated at 0 mm) to "extremely" (indicated at 100 mm). All measures are reported at area under the curve for 0 to 630 min.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: Total PFC AUC (mm*630 min)
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
Total PFC AUC (mm*630 min)
  SP-PLANT: Prospective Food Consumption | 19158 (1638) | 24889 (2060)
  SP-BEEF: Prospective Food Consumption | 19847 (1583) | 25929 (2270)
  HP-BEEF-EVEN: Prospective Food Consumption | 19087 (1537) | 21015 (1746)
  HP-BEEF-Skew: Prospective Food Consumption | 20520 (1809) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

7. Secondary Outcome: Perceived Desire to Eat
Description: Questionnaires assessing desire to eat will be completed throughout each of the 12-hour testing days (which are separated by 3-4 weeks). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The scale is 0 to 100mm. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not at all" (indicated at 0 mm) to "extremely" (indicated at 100 mm). All measures are reported at area under the curve for 0 to 630 min.
Time Frame: 5 months
Measure: Mean (Standard Error); unit: Total Desire to Eat AUC (mm*630 min)
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Number analyzed (Participants) | 17 | 17
Total Desire to Eat AUC (mm*630 min)
  SP-PLANT: Daily Desire to Eat | 18132 (1952) | 24309 (2601)
  SP-BEEF: Daily Desire to Eat | 18753 (1875) | 25886 (2566)
  HP-BEEF-EVEN: Daily Desire to Eat | 18179 (1951) | 19921 (1904)
  HP-BEEF-SKEW: Daily Desire to Eat | 19540 (1998) | NA (NA) — This group did not receive the HP-BEEF-SKEW Treatment.

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Description: Adverse event monitoring occurred throughout the study.
Arm/Group | Energy Balance Comparison | Energy Restriction Comparison
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No